CLINICAL TRIAL: NCT04883307
Title: A Randomized Trial to Investigate the Impact of Professional Development Coaching Programs in MGH Residency & Fellowship Programs, and in Women Residents in a Professional Surgical Society
Brief Title: Investigating the Impact of Professional Development Coaching Programs in Residents & Fellows
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Kerri Palamara McGrath, MD, Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2017P000569
Record Dates: First submitted 2021-04-30; First posted 2021-05-12 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Burnout, Professional
Keywords: physician burnout; physician well-being; coaching; graduate medical education; surgery
MeSH Terms: conditions — Burnout, Professional

STUDY DESIGN:
Intervention Model Description: All participants (coaches and coachees) were required to complete a baseline questionnaire including an informed consent item, demographic characteristics, Professional Fulfillment Index (PFI), Positive Emotion, Engagement, Relationship, Meaning, and Accomplishment scale (PERMA), Intolerance of Uncertainty scale (IUS), and Hardiness Resilience Score (HRS).10-13 Region was determined using self-reported cities and states as laid out in the US Census Divisions.14 Field of specialty or prospective specialty was also noted. The participating surgical residents were then randomized to the intervention group or the control group based on PFI's burnout sub-scale's quartile scores at pre-survey. Residents in the intervention group were encouraged to meet with a trained faculty coach for a 1:1 coaching meeting 3 times over 9 months. Residents in the control group were emailed wellness resources.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coaching Intervention (Experimental): Paired with a coach outside of their specific area of interest; encouraged to meet 3 times over 9 months for a 1:1 coaching meeting
  Interventions: Behavioral: Coaching
- Wellness Resources (Active Comparator): Emailed wellness resources
  Interventions: Behavioral: Wellness resources

INTERVENTIONS:
Behavioral: Coaching — Professional development coaching based on a curriculum of positive psychology principles and coaching principles.
  Arms: Coaching Intervention
Behavioral: Wellness resources — Residents in the control group received three emails across the 9 month study period that contained materials related to physician well-being such as personal development and resilience, mindfulness, and work life-integration. Materials included recommended readings, videos, and exercises and were curated by members of the Association of Women Surgeons who were not involved in the coaching program.
  Arms: Wellness Resources

SUMMARY:
The goal of the Professional Development Coaching Program is to allow trainees to understand their development over time, find meaning and purpose in their work, and identify their strengths and how to use these to overcome challenges and stressors. Additionally, the program connects trainees with a faculty member who will work with them, grow to know them in-depth over time, and provide meaningful guidance throughout the relationship. There is an additional benefit to the coaches themselves, who are able to connect with other faculty coaches in a rewarding way, that provides faculty development in leadership development and positive psychology, and space to interact with a group of like-minded physicians.

DETAILED DESCRIPTION:
A randomized controlled trial was performed to evaluate the effects of coaching on wellness, fulfillment and burnout through AWS from 2018-2020. The research protocol and all research materials and methods were reviewed and approved by the Mass General Brigham Institutional Review Board (Protocol #: 2017P00056) and funded through a grant provided by the Physicians Foundation.

AWS is a global, professional surgical society whose mission is to "to inspire, encourage, and enable women surgeons to realize their professional and personal goals."9 Concordant with its mission, the organization launched a formal coaching program in which practicing surgeons would volunteer to be trained in positive psychology coaching and paired with women surgical trainees for a remote coaching relationship.

Participants, randomization and outcome measures Members of AWS were recruited to participate in the study as coaches (attendings) or coachees (residents) via direct emails and social media. Attending surgeons were required to be women members of AWS, be in active surgical or surgical subspecialty practice and were required to reside in the United States (US) or Canada to be eligible to be a coach. Coachees were also women members of AWS, residents of the US and Canada, and were actively in residency training for the duration of the program.

All participants (coaches and coachees) were required to complete a baseline questionnaire including an informed consent item, demographic characteristics, Professional Fulfillment Index (PFI), Positive Emotion, Engagement, Relationship, Meaning, and Accomplishment scale (PERMA), Intolerance of Uncertainty scale (IUS), and Hardiness Resilience Score (HRS).10-13 Region was determined using self-reported cities and states as laid out in the US Census Divisions.14 Field of specialty or prospective specialty was also noted. The participating surgical residents were then randomized to the intervention group or the control group based on PFI's burnout sub-scale's quartile scores at pre-survey. After the 9-month study period, all participants received a follow up questionnaire similar to the baseline questionnaire. Those who completed the follow up questionnaire received a digital $10 gift card to an online shopping vendor as remuneration for study completion.

Intervention - The AWS Coaching Project Coaches who participated in the study completed a 3-hour in-person coaching training program at the 2018 and 2019 Association of Women Surgeons national meetings. Coaching materials were created by an author who is an expert in professional development coaching (K.P). in conjunction with the McLean Hospital Institute of Coaching. Training was interactive and led by Dr. Palamara and emphasized the basics principles of positive psychology and coaching. The coaches were supplied with a training manual with step by step guides for three coaching sessions with their coachees developed for this program (link to website). Each meeting was expected to be 45-60 minutes in length. In addition, coaches were also invited to participate in up to two additional optional 90-minute refresher training sessions which were offered virtually over a web-based video platform. Unique aspects of the curriculum tailored to the study population included discussion of imposter syndrome, the glass ceiling in surgery, and microaggressions. Additional details regarding the coaching training and program are published separately. 6,7 Upon completion of training, coaches were paired with 1-2 residents who were randomized to the coaching intervention group. Coach-coachee pairings were constructed based on divergent surgical specialty and geographic location to create a safe space and minimize the possibility of a more traditional mentoring relationship. All coaching sessions occurred remotely over voice or video calls. Participants were encouraged to meet for at least 3 coaching sessions over the 9-month intervention period but could meet more frequently if amenable to both parties.

Residents in the control group received three emails across the 9 month study period that contained materials related to physician well-being such as personal development and resilience, mindfulness, and work life-integration. Materials included recommended readings, videos, and exercises and were curated by members of the Association of Women Surgeons who were not involved in the coaching program.

ELIGIBILITY:
Inclusion Criteria:

* Surgical resident in the US or Canada

Exclusion Criteria:

* Surgical resident from other countries; non-surgical residents

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — This is a surgical society for female surgeons; anyone self-identifying as female can be a member.
Enrollment: 237 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2020-06-25 (Actual)

PRIMARY OUTCOMES:
Professional Fulfillment Index | Change from Baseline PFI to End of Study PFI at 9 months
  Stanford PFI
PERMA 15-item Self-scoring Instrument | Change from Baseline PERMA to End of Study PERMA at 9 months
  Positive Emotion, Engagement, Relationship, Meaning, and Accomplishment 15 item self-scoring scale (15-75); higher scores mean a better outcome

SECONDARY OUTCOMES:
Intolerance of Uncertainty | Change from Baseline IUS to End of Study IUS at 9 months
  IUS 10; higher scores mean a worse outcome
Hardiness Resilience Score | Change from Baseline HRS to End of Study HRS at 9 months
  Dispositional-resilience Scale-15; range from 0-80; higher scores mean a better outcome
Gratitude Questionnaire Six Item Form (GQ-6) | Change from Baseline gratitude to End of Study gratitude at 9 months
  GQ6; Range 6-42; higher scores mean a better outcome
Measurement of Current Status Part A | Change from Baseline coping to End of Study coping at 9 months
  MOCS Part A Questions 5-7; Range 0-12; higher scores mean a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Kerri Palamara, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
This is well-being and burnout data on surgical residents in training; sharing individual participant data may impact their career trajectory.

REFERENCES:
- [Derived] Palamara K, McKinley SK, Chu JT, Merrill AL, Yu L, Parangi S, Makowski MS, Park YS, Donelan K, Stein SL. Impact of a Virtual Professional Development Coaching Program on the Professional Fulfillment and Well-Being of Women Surgery Residents: A Randomized Controlled Trial. Ann Surg. 2023 Feb 1;277(2):188-195. doi: 10.1097/SLA.0000000000005562. Epub 2022 Jun 29. PMID 35766397

DOCUMENTS (1):
  • Study Protocol (2018-04-10): https://cdn.clinicaltrials.gov/large-docs/07/NCT04883307/Prot_000.pdf